CLINICAL TRIAL: NCT04084964
Title: NWE CHANCE Feasibility Study of a Home Hospitalisation Strategy for Patients With an Acute Episode of Heart Failure Using Integrated eHealth Applications.
Brief Title: Feasibility Study of a Home Hospitalisation Strategy for Patients With Heart Failure
Acronym: NWECHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Isala (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Professor, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NWE 661
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The NWE-Chance feasibility study is an international, multicenter, single-arm prospective and interventional study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): These patients receive the home-hospitalisation platform
  Interventions: Other: Home-hospitalisation platform for heart failure

INTERVENTIONS:
Other: Home-hospitalisation platform for heart failure — The primary objective of the INTERREG NWE-Chance project is the development of an integrated home-hospitalisation platform and the assessment of the feasibility of a home hospitalisation strategy for heart failure patients.

SUMMARY:
This feasibility study is part of a larger interregional European project (NWE-Chance) financially supported by the 'Interreg North West Europe' program to develop and validate promising integrated eHealth applications combined with nanotechnology for hospitalisation of heart failure patients at home. For more information on this research project and the partners see http://www.nweurope.eu/nwe-chance

DETAILED DESCRIPTION:
Patients participating in the NWE-Chance study will be transferred to their home supported by the integrated home hospitalisation platform and a daily visit by a specialised nurse. The home hospitalisation platform allows monitoring vital signs of patients by using the Sensium patch and a connected weighing scale and blood pressure meter of HC@home. Blood parameters like creatinine and potassium will be measured (daily) by using the Medimate lab-on-chip technology (more information below). Patients will get a smartphone to receive reminders for measurements of blood pressure and weight and will be able to see the evolution of their blood pressure and weight values. The patient application also contains educational information for the patient on home hospitalisation and on how to take the measurements correctly.

Patients are treated by a team of specialised nurses under supervision of a cardiologist. The nurses visit patients at least once a day and are equipped with laboratory equipment and IV medication administering equipment. These devices and equipment are currently used in standard HF care and are not part of the newly developed home hospitalisation platform. Patients receive treatment similar to in-hospital treatment, according to the cardiologist's best knowledge and insight.

In the case of Jessa Hospital, if there would be a need for IV medication during the home-hospitalisation period, this will lead to rehospitalisation of the patient and the ending of the intervention. In Isala, the nurses have a 24/7 duty service and can be called by patients or their relatives on their own initiative. In Jessa hospital and MUMC+, the nursing team can be contacted between 9 AM and 17 PM. During other hours, the patients can contact the cardiologist on call.

In case of treatment failure or severe deterioration, patients will be transported to the hospital. In case of emergency, ambulances will transport patients to the hospital (conversion to regular hospitalisation). If in follow-up, condition worsens, the patient can be readmitted at home again. In theory, patients may undergo repeated hospitalisations at home.

The home-hospitalisation period will last at least 5 days and can be extended, till a maximum of 13 days, after consultation of a cardiologist. Patient will be asked to fill in questionnaires to assess feasibility at the end of the home-hospitalisation period (last visit of nurse). At the last visit of the nurse, she will take all the devices with her.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known and well assessed chronic heart failure.
* Age>18 years
* (Indication for) hospital admission for acute decompensated heart failure
* Living within a wide proximity of the hospital (differs per centre)
* Living independently and/or sufficiently supported at home and/or living in nursing homes (or other supported living modalities).

Exclusion Criteria:

* Indication for IC/CCU admission;
* Contraindication to Chance@Home;
* Mental impairment leading to inability to cooperate;
* Severe comorbidity requiring simultaneous hospital care;
* History of severe liver / kidney disease;
* Unstable blood pressure (systolic blood pressure <90mmHg);
* Unstable heart rhythm (in case of sinus rhythm, heart rate >110/min, in case of atrial fibrillation >150/min);
* Need for intravenous inotropic medication;
* Unstable respiratory condition (sO2 <90% without additional O2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability will be assessed with the SUTAQ questionnaire adapted for home-hospitalisation | 5-14 days
  The SUTAQ or the Service User Technology Acceptability Questionnaire is to measure acceptability and identify the characteristics of persons who were likely to reject technological health services Will be assessed after the home-hospitalisation in patients and staff. There are 20 questions that can be answered with 6 answer possibilities ranging from fully disagree to fully agree. These answered will be coded to numbers ranging from 1-6 (6 is fully agree, 1 fully disagree). The total score is 120 and the range for the score can be 20-120
Usability will be assessed with the SUS questionnaire adapted for home-hospitalisation | 5-14 days
  SUS or the System Usability Scale will be used after the home-hospitalisation to assess the usability of the platform for the patients and staff. There are 10 questions in total with 5 answer possibilities ranging from totally agree to fully disagree. The answers will be coded to numbers (1-5) and 5 means totally agree and 1 is fully disagree. The total score is 50 and the range for the score can be 10-50
Satisfaction will be assessed with the Satisfaction Home-hospitalisation program questionnaire | 5-14 days
  The satisfaction of the home-hospitalisation program questionnaire consist of 19 questions and will be used to assess the satisfaction of patients. There are 5 answer possibilities ranging from completely satisfied to very dissatisfied. The answers will be coded to numbers (1-5) and 5 means completely satisfied and 1 is very dissatisfied. The total score is 95 and the range for the score can be 19-95
Platform use will be assessed with the amount of logs in the patient application | 5-14 days
Number of adverse events will be mapped by the study team | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leenen JPL, Scherrenberg M, Bruins W, Boyne J, Vranken J, Brunner la Rocca HP, Dendale P, van der Velde AE. Usability of a digital health platform to support home hospitalization in heart failure patients: a multicentre feasibility study among healthcare professionals. Eur J Cardiovasc Nurs. 2024 Mar 12;23(2):188-196. doi: 10.1093/eurjcn/zvad059. PMID 37294588